CLINICAL TRIAL: NCT02352701
Title: Efficacy and Safety of Basic Triple Therapy Including Ilaprazole, Levofloxacin on the First Line Eradication Treatment of H.Pylori
Brief Title: Efficacy and Safety of Basic Triple Therapy Including Ilaprazole on the First Line Eradication Treatment of H.Pylori
Status: Completed | Type: Observational
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CMC-LDS-ILA01
Record Dates: First submitted 2015-01-26; First posted 2015-02-02 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Helicobacter Infections
Keywords: helicobacter pylori; ilaprazole; eradication; triple therapy
MeSH Terms: conditions — Helicobacter Infections | interventions — ilaprazole; Amoxicillin; Levofloxacin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Noltec®,ChongkundangAmoxicillin®,Cravit®: Noltec tab 10mg, Chongkundang Amoxicillin Cap 500mg 2caps and Cravit tab 500mg by oral, twice a day for 10 days
  Interventions: Drug: Noltec tab. 10mg; Drug: Chongkundang Amoxicillin Cap. 500mg; Drug: Cravit Tab. 500mg

INTERVENTIONS:
Drug: Noltec tab. 10mg — Ilaprazole 10mg BID dosage form : delayed release tablet
  Other Names: Ilaprazole
Drug: Chongkundang Amoxicillin Cap. 500mg — Amoxicillin 1000mg, BID dosage form : capsule
  Other Names: Amoxicillin
Drug: Cravit Tab. 500mg — Levofloxacin 500mg, BID dosage form : film coated tablet
  Other Names: Levofloxacin

SUMMARY:
This study compared efficacy and safety of basic triple therapy including Ilaprazole 10mg, Levofloxacin 500mg and Amoxicillin 1000mg BID for 10 days on the first line eradication treatment of H.pylori

DETAILED DESCRIPTION:
This study compared efficacy and safety of basic triple therapy including Noltec(Ilaprazole) 10mg, Cravit(Levofloxacin) 500mg and Chongkundang Amoxicillin Cap(Amoxicillin) 1000mg BID on the first line eradication treatment of H.pylori.

Participants are defined as persons who have endoscopically confirmed on gastric or duodenal ulcer(including scar stage) and gastritis confirmed to be H.pylori positive patients in the biopsy and UBT test. For 10 days, Participants treated as basic triple therapy including Noltec(Ilaprazole) 10mg, Cravit(Levofloxacin) 500mg and Chongkundang Amoxicillin Cap(Amoxicillin) 1000mg BID. After treatment, The healing rate was evaluated in the UBT test and Biopsy at 49±5days from the first day dosing.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have endoscopically confirmed on gastric, duodenal ulcer(including scar) or gastritis confirmed to be H.pylori positive patients in the biopsy and UBT test.
* Subject who fully understands conditions of clinical trial.
* Subject who agrees to participate and spontaneously sign the ICF

Exclusion Criteria:

* Known hypersensitivity to any component of ilaprazole, Amoxicillin and Levofloxacin
* Subjects who are taking contraindicated medications for experimental and concomitant drug.
* Patients with abnormal levels in the laboratory tests

  * Total Bilirubin, Creatinine> 1.5 times upper limit of normal
  * AST, ALT, Alkaline phosphatase, BUN> 2 times upper limit of normal
* Administrated of PPI, antibiotic medication within 4 weeks prior to commencement of the study.
* Pregnant and/or lactating women
* Reproductive aged women not using contraception
* Uncontrolled diabetics
* Uncontrolled hypertension
* Uncontrolled liver dysfunction
* Alcoholics
* Subjects with a history of digestive malignancy within 5 years
* Subjects with a history of gastrectomy or esophagectomy
* Subjects with hereditary diseases such as Galactose intolerance, Lapp lactose deficiency, glucose-galactose malabsorption.
* Subjects participating in a clinical trial before another trial wihin 30 days
* Inconsistence judged subject by researcher

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited the hospital
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The eradication rate of H.pylori at Day 49±5 as assessed by UBT test and Biopsy | Day 49±5
  The eradication rate of H.pylori after 10 days treatment is defined as those participants who have endoscopically confirmed on gastric or duodenal ulcer(including scar stage) and gastritis confirmed to be H.pylori positive patients in the biopsy and UBT test.
  The treatment : Noltec(Ilaprazole) 10mg+Chongkundang Amoxicillin(Amoxicillin) 1000mg+Cravit(Levofloxacin) 500mg was administered twice a day for 10days

SECONDARY OUTCOMES:
The safety of Noltec(Ilaprazole) 10mg BID treatment at Day 49±5. Record the number of patients with adverse Events | Day 49±5
  Record the number of patients with adverse Events. Also Record the symptoms, date, duration, and intensity of Adverse events such.
The healing rate of gastritis and ulcers at Day 49±5 as assessed by endoscopy confirmed to be active stage, healing stage and scarring stage. | Day 49±5
The rate of patients with Clarithromycin resistance as assessed by biopsy after treatment. | Day 49±5

CONTACTS AND LOCATIONS:
Overall Officials: Dongsoo Lee, MD, PhD., Principal Investigator — The Catholic Univ. of Korea, Daejeon St.Mary Hospital
Locations (1):
- The Catholic Univ. of Korea Daejeon St.Mary Hospital, Daejeon, South Korea